CLINICAL TRIAL: NCT03653039
Title: Sammenligning Mellem Standard Tube og Den Ultra-tynde Tritube® Til Intubation, og Til Opretholdelse af Adgang Til Trachea Efter anæstesi, Hos Patienter Med Forventet Vanskelig Direkte Laryngoskopi
Brief Title: Comparison Between a Standard Tube and the Ultra-thin Tritube for Intubation of the Trachea and for Maintaining Access to the Trachea After Anaesthesia, in Patients With an Expected Difficult Direct Laryngoscopy
Acronym: Tritube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Seltz Kristensen (Other)
Responsible Party: Sponsor-Investigator, Michael Seltz Kristensen, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-18023689 Tritube
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Oral Neoplasm; Pharynx Cancer; Larynx Cancer
MeSH Terms: conditions — Mouth Neoplasms; Pharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tritube (Experimental)
  Interventions: Device: Tritube
- Standard endotracheal tube (Active Comparator)
  Interventions: Device: Standard enditracheal tube

INTERVENTIONS:
Device: Tritube — The ultra thin tribute is used used for the ventilation of the patients in this arm
  Arms: Tritube
Device: Standard enditracheal tube — A standard endotracheal tube is used used for the ventilation of the patients in this arm
  Arms: Standard endotracheal tube

SUMMARY:
The investigators compare the ease of intubation between a new ultra-thin endotracheal tube, "Tritube", and a standard endotracheal tube in patients with predictors of difficult laryngoscopy. Furthermore the investigators compare the acceptance of leaving the Tritube in trachea after end of anaesthesia, with the use of a tube exchange catheter.

DETAILED DESCRIPTION:
In patients scheduled for surgery and anaesthesia in the Head-/neck/ear/nose/throat -region the investigators compare the ease of tracheal intubation between a new ultra-thin endotracheal tube, "Tritube", and a standard endotracheal tube in patients with predictors of difficult laryngoscopy. The intubation is performed with an angulated video laryngoscope.

Furthermore the investigators compare the acceptance of leaving the Tritube in trachea after end of anaesthesia, with the use of a tube exchange catheter. The latter continues into the post-operative recovery-ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients for anaesthesia for surgery in the Head-/neck/ear/nose/throat
* planned for oral intubation with video-laryngoscopy
* with risk factors for difficult direct laryngoscopy

Exclusion Criteria:

* Patient with increased secretions in the airway (Pneumonia, bronchitis, productive cough)
* Patients planned for awake intubation
* Patients where mask-ventilation is judged to could become impossible
* Patients where access to the cricothyroid membrane is judged to be difficult or impossible
* Patients in ASA (american Society of Anaesthesiologists) physical classification status >3
* Patients who are scheduled for rapid sequence induction (RSI) due to risk of aspiration
* Patients with stridor
* Patients with hypoxemia (Saturation < 90 % in room air)
* Operation duration planned to > 2.5 hours
* Patients with the need for a nerve-stimulation-tube during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Rate of Excellent intubation conditions | 2 hours
  Rate of Excellent intubation conditions judged on the scale excellent/good/fair/poor

SECONDARY OUTCOMES:
The rate of interruption by the tube of the view to the vocal cords at any time, to such a degree that it disturbs the intubation | 2 hours
The Intubation Difficulty Score (IDS) | 2 hours
  The intubation difficulty scale , range 0 to 7, 0 indicates easy intubation, 1 - 5 indicates slight difficulty, 5< indicates moderate to major difficulty
Time to intubated | 2 hours
  Time from the tube is advanced past the vocal cords until the cuff is inflated in the trachea
Time to the patient becomes ventilated via the tube | 2 hours
  Time from the tube is advanced past the vocal cords until the cuff is inflated in the trachea and CO2 waveform is observed
Number of intubation attempts | 2 hours
  one attempt is every-time the tube is advanced past the incisors
The rate of succesful intubation with 60 seconds | 1 minute
Number of remodellings of the stilette | 2 hours
rate of use for "reverse loading" of the tube on the stylet | 2 hours
the "percent of glottic opening" , (POGO), Before the tube is inserted | 2 hours
the"percent of glottic opening" , POGO, with the tube in place | 2 hors
Intubation conditions Strom scale | 2 hours
  Direction of the tube-stylet combination excellent/good/poor, easy/fair/difficult. Advancement of the tube-stylet combination excellent/good/poor easy/fair/difficult
The surgeons score of the space and working conditions in the mouth/pharynx and larynx after intubation | 2 hours
The difference between ET CO2 and arterial blood-gas CO2 after 15 minutes of surgery | 20 minutes
the duration of the Tritube being in the trachea after return of spontaneous ventilation and deflation of the cuff /(Tritube group) | 4 hours
The duration of the tube-exchange catheter being in the trachea after its placement / (Tube-exchange-catheter group) | 4 hours
The ration of patients who still has the Tritube or the tube-exchange-catheter in place when arriving in the post-operative recovery unit | 4 hours
The ration of patients who still has the Tritube or the tube-exchange-catheter in place one hour after arrival in the Post anaesthesia care unit the post-operative recovery unit | 4 hours
The patient's satisfaction with having the Tritube or the tube-exchange-catheter in place when being awake in the Post anaesthesia care unit | 4 hours
  Visual analog scale from 1-10, 1= no nuisance, 10= unberable

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kristensen, MD, Principal Investigator — Rigshospitalet, University Hospital of Copenhagen Denmark
Locations (1):
- Rigshospitalet, section for anaesthesia for ENT and Maxillofacial surgery, section 3071, Copenhagen, Denmark

REFERENCES:
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Kristensen MS, de Wolf MWP, Rasmussen LS. Ventilation via the 2.4 mm internal diameter Tritube(R) with cuff - new possibilities in airway management. Acta Anaesthesiol Scand. 2017 Jul;61(6):580-589. doi: 10.1111/aas.12894. Epub 2017 Apr 23. PMID 28436022
- [Background] Strom C, Barnung S, Kristensen MS, Bottger M, Tvede MF, Rasmussen LS. Tracheal intubation in patients with anticipated difficult airway using Boedeker intubation forceps and McGrath videolaryngoscope. Acta Anaesthesiol Scand. 2015 Oct;59(9):1154-60. doi: 10.1111/aas.12543. Epub 2015 May 16. PMID 25982220